CLINICAL TRIAL: NCT04604431
Title: Intervention to Reduce Early (Peanut) Allergy in Children
Acronym: iREACH
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Ruchi S Gupta, Professor, Ann & Robert H Lurie Children's Hospital of Chicago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AAABB-U01-LCH-00; U01AI138907 (NIH)
Record Dates: First submitted 2020-10-14; First posted 2020-10-27 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Food Allergy Peanut; Food Allergy in Infants
Keywords: Food Allergy; Peanut Allergy Incidence; Clinical Decision Support Tool; Infants; Peanut Allergy Prevention
MeSH Terms: conditions — Peanut Hypersensitivity; Food Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (CDS Tool Integrated) (Experimental): Pediatric clinicians in this arm will receive the iREACH CDS tool and education on the PPA Guidelines to support adherence to the Guidelines.
  Interventions: Other: iREACH CDS Tool
- Control (No CDS Tool Integrated) (No Intervention): No study procedures will be implemented in the control practices, and their pediatric clinicians will not receive extra PPA Guidelines education, nor will any EHR modifications be made in their practices to support adherence to PPA Guidelines.

INTERVENTIONS:
Other: iREACH CDS Tool — Pediatric clinicians in the intervention arm will 1) receive the iREACH education module, 2) have the iREACH CDS tool integrated into the EHR templates for use at the 4-, 6-, 9-, 12-month WCC, and 3) will be reminded by EHR-embedded prompts at the 9-month WCC to ask caregivers whether peanuts were introduced and tolerated.
  Arms: Intervention (CDS Tool Integrated)

SUMMARY:
iREACH is a five-year NIH funded study aimed at assessing and improving pediatric clinician adherence to the 2017 NIAID Prevention of Peanut Allergy (PPA) Guidelines.

iREACH has been developed as an electronic health record (EHR) integrated Clinical Decision Support (CDS) tool together with educational modules on the PPA guidelines to assist clinicians in implementing the 2017 NIAID PPA Guidelines.

A practice-based, two-arm, cluster-randomized clinical trial will evaluate the effectiveness of iREACH in increasing pediatric clinician adherence to the PPA Guidelines and explore the end-goal of reducing peanut allergy incidence by age 2.5 years in the intervention vs control group.

This study has the potential to: 1) provide evidence regarding the effectiveness of iREACH in promoting clinical processes and outcomes related to the PPA Guidelines, 2) provide important insight about practice-based implementation of PPA Guidelines by pediatric clinicians, allergists and caregivers, and 3) facilitate rapid, widespread implementation of PPA Guidelines and reduce peanut allergy incidence across the US.

DETAILED DESCRIPTION:
A minimum of 30 pediatric practice sites will be randomized to the iREACH intervention arm or to the control arm.

Primary Objective To determine the effectiveness of iREACH in increasing adherence to the PPA Guidelines among pediatric clinicians.

Secondary Objective To determine the effectiveness of iREACH in decreasing the incidence of peanut allergy by age 2.5.

Exploratory Objectives

1. To determine allergists' adherence to the PPA Guidelines
2. To identify common barriers/facilitators for PPA Guideline adherence among pediatric clinicians and caregivers
3. To determine caregiver adherence to the PPA Guidelines

All pediatric clinicians within each participating practice (n≈200 total) will be assigned to the arm to which their practice is randomized. The trial will be conducted over an 18-month period. During this time, approximately 500 high-risk infants and 10,000 low-risk infants are expected to be seen for 4- and 6-month well child care visit (WCC). The primary outcome, pediatric clinician adherence to the PPA Guidelines, will be assessed using EHR data for each infant following the 6-month WCC.

Data for the secondary outcome will be obtained by a combination of EHR data extracted after the infant's 6-month WCC and data collected from caregivers. EHR data extraction will be performed to obtain data from the infant's 9-, 12-, 15-, 18-, 24-month WCC and any sick visits and allergist progress notes entered from 4-30 months of age. Caregivers' data will be collected via surveys of caregivers of children seen for 4- or 6-month WCC visits during the study period. Caregivers will be recruited and asked to provide informed consent at the time of the child's first birthday and questions will be asked to determine the incidence of peanut allergy. A follow-up survey will be sent to caregivers after the child's second birthday.

Data for exploratory outcomes will be obtained through EHR data extraction and surveys of pediatric clinicians and the caregivers of infants seen for 4- or 6-month WCC. Pediatric clinicians in the intervention arm will be asked to provide informed consent and will complete three surveys over approximately 21 months. Pediatric clinicians in the control arm will be asked to provide informed consent following completion of data collection for the primary outcome and will complete one survey. Finally, caregivers, through the two surveys conducted at the time of their child's first and second birthdays, will provide information for exploratory outcomes.

ELIGIBILITY:
Inclusion Criteria:

Practice sites

* The practice utilizes a centrally-integrated EHR.
* The practice has signed a legally-binding engagement agreement with Lurie Children's Pediatric Practice Research Group.
* The practice employs at least one physician who has completed a residency in general pediatrics and is practicing as a general pediatrician.

Pediatric Clinicians:

* Clinician is a physician, physician assistant, resident, advanced practice nurse, family practitioner, or pediatric nurse practitioner working in a pediatric practice.
* Clinician is employed by a practice that is a member of one of the participating practices in the study.
* Clinician provides well child care to infants ages 4 or 6 months.

Infants • Infant has been seen by a pediatric clinician in the intervention or control arm for a 4- and/or 6-month WCC.

Caregivers

* Is the caregiver of an infant seen for a 4- and/or 6-month WCC by a pediatric clinician in a practice belonging to the study's intervention or control arms.
* Is 18+ years of age or has parent or guardian permission to participate.
* Is able to understand the study and provide informed consent for the 12- and 24-month (child's age) survey.

Exclusion Criteria:

Practice Sites

* Sees <50 newborn patients/year.
* Has only temporary pediatricians on staff.
* The practice pediatric clinicians do not use an EHR system.

Pediatric clinicians

* The clinician is a temporary employee.
* The clinician begins employment at participating practice less than three months prior to end of the 18-month study enrollment period.

Infants

* The infant has a medical condition that chronically inhibits the ability to take food orally (i.e., dysphagia, muscular dystrophy, gastrostomy).
* The infant has past or current medical problems or findings from physical examination or laboratory testing not listed above for which the pediatric clinician indicates that implementation of PPA Guidelines may pose a medical risk other than allergic reactions or may interfere with the infant's appropriate implementation of the PPA Guidelines or study investigators conclude that implementation of the PPA Guidelines was not possible or may have impacted the quality or interpretation of the data obtained from the study.

Caregivers

• Caregiver's primary language is not English or Spanish.

Min Age: 4 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-11-04 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2025-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Ruchi S Gupta, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (30):
- United States (30):
  - Pediatric Associates of Arlington Heights, SC-PEDIATRUST, Arlington Heights, Illinois
  - OSF Medical Group Pediatrics Bloomington, Bloomington, Illinois
  - Child and Adolescent Health Associates, Chicago, Illinois
  - Northwestern Children's Practice, Chicago, Illinois
  - Streeterville Pediatrics, Chicago, Illinois
  - Erie Family Health Centers - Erie Teen and Young Adult Health Center, Chicago, Illinois
  - Erie Family Health Centers - West Town, Chicago, Illinois
  - Erie Family Health Centers - Helping Hands - Foster, Chicago, Illinois
  - Lurie Children's Primary Care Town & Country Pediatrics, Chicago, Illinois
  - Near North Health Services Corporation, Chicago, Illinois
  - Children's Health Associates, Chicago, Illinois
  - Lakeview Pediatrics, Chicago, Illinois
  - OSF Medical Group Pediatrics Danville, Danville, Illinois
  - Erie Family Health Centers - Evanston, Evanston, Illinois
  - Lurie Children's Primary Care Chicago Area Pediatrics, Evanston, Illinois
  - OSF Medical Group Pediatrics Godfrey, Godfrey, Illinois
  - Pediatric Partners, SC-PEDIATRUST, Highland Park, Illinois
  - Bedrose Pediatrics, Hoffman Estates, Illinois
  - Lake Shore Pediatrics, SC-PEDIATRUST, Libertyville, Illinois
  - OSF Medical Group (MG)-Morton Pediatrics, Morton, Illinois
  - Ad-Park Pediatrics, SC-PEDIATRUST, Northbrook, Illinois
  - Oak Park Pediatrics, Oak Park, Illinois
  - University of Illinois College of Medicine Peoria, Peoria, Illinois
  - OSF-Center for Health (CFH)-Route 91, Peoria, Illinois
  - Woodfield Pediatrics, SC-PEDIATRUST, Schaumburg, Illinois
  - OSF Medical Group (MG) Washington, Washington, Illinois
  - Erie Family Health Centers - Waukegan, Waukegan, Illinois
  - Wheaton Pediatrics, SC-PEDIATRUST, Wheaton, Illinois
  - Pediatric Associates of the North Shore, Wilmette, Illinois
  - Elm Street Pediatrics, SC-PEDIATRUST, Winnetka, Illinois

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bilaver LA, Ariza AJ, Binns HJ, Jiang J, Cohn R, Sansweet S, Hultquist H, Panza JL, Togias A, Gupta RS. Design of the Intervention to Reduce Early Peanut Allergy in Children (iREACH): A practice-based clinical trial. Pediatr Allergy Immunol. 2024 Apr;35(4):e14115. doi: 10.1111/pai.14115. PMID 38566365
- [Background] Samady W, Negris O, Jiang J, Bilaver LA, Gupta RS. Developing an infant atopic dermatitis scorecard for pediatric clinicians. Ann Allergy Asthma Immunol. 2024 Oct;133(4):469-470. doi: 10.1016/j.anai.2024.06.009. Epub 2024 Jun 15. No abstract available. PMID 38880210
- [Result] Samady W, Bilaver LA, Jiang J, Iyer A, Laurienzo Panza J, Togias A, Gupta RS. Evaluation of Training to Increase Knowledge of the Addendum Guidelines for the Prevention of Peanut Allergy in the US. JAMA Netw Open. 2023 Mar 1;6(3):e234706. doi: 10.1001/jamanetworkopen.2023.4706. PMID 36961467

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participating practices (n=30) were recruited and enrolled prior to the start of the study. During an 18-month observation period (start date varied by network), 290 clinicians and 18480 infants seen for 4- and/or 6- month well child care visits were observed via electronic health records (EHR). EHR notes were pulled between November 1, 2020 through October 31, 2022. EHR data was available for use per the agreements outlined during practice recruitment.
Pre-assignment Details: For the primary outcome, practices were enrolled and randomized. No individual participants were enrolled. 37 practices were invited. 7 practices decided not to participate. Finally, 30 practices were enrolled and randomized into the intervention vs control arm based off of annual patient volume of 4- and 6-month well child care (WCC) visits. Four patient volume strata were considered (<500 visits, 500-999, 1000-1499, ≥1500). Practices were randomized in a 1:1 ratio within each stratum.
Units Other Than Participants: practices
Groups:
- Intervention (CDS Tool Integrated): Pediatric clinicians in all intervention practices received the iREACH clinical decision support (CDS) tool and education on the Prevention of Peanut Allergy (PPA) Guidelines to support adherence to the Guidelines. All infants in the intervention arm were observed.
  iREACH CDS Tool: Pediatric clinicians in the intervention arm will 1) receive the iREACH education module, 2) have the iREACH CDS tool integrated into the EHR templates for use at the 4-, 6-, 9-, 12-month WCC, and 3) will be reminded by EHR-embedded prompts at the 9-month WCC to ask caregivers whether peanuts were introduced and tolerated.
Period: Overall Study
Arm/Group | Intervention (CDS Tool Integrated) | Control (No CDS Tool Integrated)
Started (Total number of clinicians and infants observed as part of the trial.) | 9476; 16 practices | 9294; 14 practices
Clinicians Observed | 186; 16 practices | 104; 14 practices
Infants Observed | 9290; 16 practices | 9190; 14 practices
Completed (Total number of clinicians and infants observed as part of the trial.) | 9476; 16 practices | 9294; 14 practices
Not Completed | 0; 0 practices | 0; 0 practices

BASELINE CHARACTERISTICS:
Population: All infants seen for a 4- and/or 6 month well child visit during an 18 month observation period were included in the analyses.
  For the primary outcome, only data relevant to the infants are reported. Clinician and parent/caregiver data are exploratory outcomes and will not yet be reported.
Groups:
- Intervention (CDS Tool Integrated): Pediatric clinicians in all intervention practices received the iREACH CDS tool and education on the PPA Guidelines to support adherence to the Guidelines. All infants in the intervention arm were observed.
  iREACH CDS Tool: Pediatric clinicians in the intervention arm will 1) receive the iREACH education module, 2) have the iREACH CDS tool integrated into the EHR templates for use at the 4-, 6-, 9-, 12-month WCC, and 3) will be reminded by EHR-embedded prompts at the 9-month WCC to ask caregivers whether peanuts were introduced and tolerated.
- Total: Total of all reporting groups
Arm/Group | Intervention (CDS Tool Integrated) | Control (No CDS Tool Integrated) | Total
Number analyzed (Participants) | 9290 | 9190 | 18480
Age, Customized [Median (Inter-Quartile Range); unit: Days]
  Age in Days | 127 [123 to 143] | 126 [123 to 141] | 126 [123 to 141]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4774 | 4692 | 9466
  Male | 4516 | 4498 | 9014
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1907 | 1082 | 2989
  Not Hispanic or Latino | 6029 | 6252 | 12281
  Unknown or Not Reported | 1354 | 1856 | 3210
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 49 | 26 | 75
  Asian | 615 | 590 | 1205
  Native Hawaiian or Other Pacific Islander | 13 | 3 | 16
  Black or African American | 580 | 926 | 1506
  White | 6139 | 5271 | 11410
  More than one race | 323 | 465 | 788
  Unknown or Not Reported | 1571 | 1909 | 3480
Region of Enrollment [Number; unit: participants]
  United States | 9290 | 9190 | 18480
Health Insurance Type [Count of Participants; unit: Participants]
  Private | 6673 | 6828 | 13501
  Public | 2359 | 1320 | 3679
  Other | 195 | 962 | 1157
  Missing | 63 | 80 | 143
Egg Allergy [Count of Participants; unit: Participants]
  Egg Allergy | 59 | 14 | 73
  No Egg Allergy | 9231 | 9176 | 18407
Eczema [Count of Participants; unit: Participants]
  Mild-Moderate Eczema | 731 | 435 | 1166
  Severe Eczema | 173 | 53 | 226
  No Eczema | 8386 | 8702 | 17088
Well Child Visits [Count of Participants; unit: Participants]
  Only 4 Month Well Child Visits | 1706 | 1449 | 3155
  Only 6 Month Well Child Visits | 1809 | 1633 | 3442
  Both | 5775 | 6108 | 11883

OUTCOME MEASURES:

1. Primary Outcome: Pediatric Clinician Adherence to Guidelines
Description: The primary endpoint is the percentage of infants within each trial arm whose pediatric clinician adhered to the guidelines regarding peanut introduction assessed after completion of either a 4- or 6-month WCC. The primary endpoint concerns only the peanut introduction recommendation by the treating pediatric clinician and not additional behavior by the treating allergist or by caregivers. The primary endpoint will be measured separately by risk category as follows:
  * % of infants at low risk for peanut allergy whose pediatric clinician adhered to the guidelines for that infant.
  * % of infants at high risk for peanut allergy whose pediatric clinician adhered to the guidelines for that infant.
Time Frame: 18 months
Population: Infants seen for a 4- and/or 6- month WCC visits. Low-risk infants (n=18182) were categorized as those with no/mild/moderate eczema and no egg allergy. High-risk infants (n=298) were categorized as those with severe eczema and/or egg allergy. Clinician adherence was analyzed with infants as the unit of analysis. Odds ratios reported
Measure: Number; unit: infants
Arm/Group | Intervention (CDS Tool Integrated) | Control (No CDS Tool Integrated)
Number analyzed (Participants) | 9290 | 9190
infants
  Adherent Low-Risk: number analyzed (Participants) | 9059 | 9123
  Adherent Low-Risk | 7607 | 3231
  Adherent High-Risk: number analyzed (Participants) | 231 | 67
  Adherent High-Risk | 62 | 7
Statistical Analysis 1: Comparison: Intervention (CDS Tool Integrated) vs Control (No CDS Tool Integrated); Odds ratios will be computed to describe the odds of adherence for the iREACH intervention compared to the control intervention for low-risk infants; Test type: Superiority; p < 0.001, Mixed Models Analysis; Odds Ratio (OR) = 14.1, 95% CI 2-sided [6.9 to 29.1]
Statistical Analysis 2: Comparison: Intervention (CDS Tool Integrated) vs Control (No CDS Tool Integrated); Odds ratios will be computed to describe the odds of adherence for the iREACH intervention compared to the control intervention for high-risk infants; Test type: Superiority; p = 0.034, Mixed Models Analysis; Odds Ratio (OR) = 3.1, 95% CI 2-sided [1.1 to 8.8]

2. Secondary Outcome: Incidence of Peanut Allergy by Age 2.5
Description: The secondary endpoint is the incidence of peanut allergy by age 2.5 years and is assessed through a combination of parent survey data and extracted EHR data. Secondary endpoints will be measured separately by risk category as follows:
  * % of infants at low risk for peanut allergy who developed peanut allergy by age 2.5.
  * % of infants at high risk for peanut allergy who developed peanut allergy by age 2.5.
Time Frame: 2 years
Reporting Status: Not Posted

3. Other Pre Specified Outcome: Allergist Adherence to the Guidelines
Description: Recommendations provided to caregiver for infant peanut product introduction.
Time Frame: 18 months
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Barriers/Facilitators to Guideline Adherence Among Pediatric Clinicians and Caregivers.
Description: What factors serve as barriers and facilitators for clinicians and caregivers to adhere to guidelines.
Time Frame: 12 to 18 months
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Caregiver Adherence to the Guidelines
Description: Whether or not caregivers follow recommendations provided by clinicians - infant peanut product introduction and feeding frequency
Time Frame: 12 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Description: No adverse events (AEs) among infants, caregivers, and pediatric clinicians were expected because this is an educational intervention trial aiming to to improve the implementation of the Prevention of Peanut Allergy Guidelines which are now considered standard of care in the USA. The intervention included education, clinical decision support tools, and supplementary aids. Therefore, AEs were not monitored/assessed.
Arm/Group | Intervention (CDS Tool Integrated) | Control (No CDS Tool Integrated)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-27): https://cdn.clinicaltrials.gov/large-docs/31/NCT04604431/Prot_SAP_000.pdf